CLINICAL TRIAL: NCT04918784
Title: Assessment of Wound Closure Comparing Synthetic Hybrid-Scale Fiber Matrix With Standard of Care in Treating Diabetic Foot Ulcer
Brief Title: Comparing Synthetic Hybrid-Scale Fiber Matrix With Standard of Care in Treating Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acera Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-RES-002
Record Dates: First submitted 2021-05-12; First posted 2021-06-09 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Synthetic Hybrid-Scale Fiber Matrix; Diabetic Foot Ulcer; Epithelialization
MeSH Terms: conditions — Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will remain blinded to the randomization assignment from the time of randomization assignment to the end of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment with Synthetic Hybrid-Scale Fiber Matrix (Experimental): Diabetic foot ulcers will be treated by application of the Synthetic Hybrid-Scale Fiber Matrix. The synthetic matrix will be applied weekly or as needed based on the clinician discretion and ongoing wound assessment.
  Interventions: Device: Restrata®
- Treatment with Standard of Care (Active Comparator): Diabetic foot ulcers will be treated by application of an appropriate dressing (foam or alginate dressing) to maintain wound moisture balance in the wound and changed daily.
  Interventions: Device: Wound Dressing

INTERVENTIONS:
Device: Restrata® — Restrata® is a sterile, single use device intended for use in local management of wounds. Restrata® is a soft, white, conformable, non-friable, absorbable matrix that provides a moist environment for the body's natural healing process to occur. Restrata® is made from synthetic biocompatible materials and was designed to include a fibrous structure with high porosity, similar to native extracellular matrix.
  Other Names: Synthetic Hybrid-Scale Fiber Matrix
  Arms: Treatment with Synthetic Hybrid-Scale Fiber Matrix
Device: Wound Dressing — Alginate or Foam wound dressing is intended to manage wounds.
  Arms: Treatment with Standard of Care

SUMMARY:
The purpose of the following prospective, randomized, controlled clinical trial is to compare synthetic hybrid-scale fiber matrix (Restrata®, Acera Surgical, Inc.) with standard of care in treating diabetic foot ulcers in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old
2. Patient is willing and capable of complying with all protocol requirements
3. Patient or legally authorized representative (LAR) is willing to provide written informed consent prior to or at the beginning of the run-in period
4. Patient has Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per American Diabetes Association)
5. Ulcer must be located at least in part on the foot or ankle
6. Ulcer must be present for a minimum of 28 days prior to randomization and initial application of study product
7. Wound size must be < 30cm2 on the day of randomization and initial application of the study product, after initial debridement
8. Patient has adequate circulation to the affected extremity, as demonstrated by at least ONE of the following within 60 days prior to enrollment/randomization:

   1. Dorsum transcutaneous oxygen test (TcPO2) of study leg with results ≥40mmHg, OR
   2. Ankle-Brachial Index (ABI) of study leg with results of ≥ 0.7
   3. Toe-Brachial Index (TBI) of study extremity with results of > 50 mmHg

Exclusion Criteria:

1. Patient has been previously enrolled into this study, or is currently participating in another drug or device study that has not reached its primary endpoint
2. Patient is pregnant, breast feeding or planning to become pregnant
3. Patient has a known allergy to resorbable suture materials, e.g. Polyglactin 910 (PGLA), Polydioxanone (PDS)
4. Patient has a life expectancy less than six months as assessed by the investigator
5. Patient has received skin substitutes during the run-in period or within 14 days prior to beginning of run-in period
6. Patient has an additional wound within 3 cm of the study wound
7. Hgb A1c > 12% within 3 months prior to randomization in patients with a known history of diabetes
8. Patient not in reasonable metabolic control in the judgment of the investigator
9. Patient with a known history of poor compliance with medical treatments
10. Patient currently undergoing cancer treatment
11. Patient has been diagnosed with at least one of the following autoimmune connective tissue diseases: lupus, vasculitis, sickle cell, or uncontrolled rheumatoid arthritis
12. Patient is taking parenteral corticosteroids or any cytotoxic agents for 7 consecutive days during the run-in period or up to 30 days before the run-in period. Chronic oral steroid use is not excluded if dose is < 10 mg per day for prednisone.
13. Active infection, undrained abscess, or critical colonization of the wound with bacteria in the judgment of the investigator
14. Osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence
15. Patient unwilling to or unable to safely utilize appropriate offloading device to unweight wound
16. Study ulcer spontaneously closes during the 2-week run in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Husain, DPM, Principal Investigator — Midwest Foot & Ankle Clinics
Locations (1):
- Midwest Foot and Ankle Clinics, Hoffman Estates, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is a 2 week run-in period to confirm eligibility prior to treatment on study
Period: Overall Study
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care
Started | 25 | 21
Completed | 19 | 18
Not Completed | 6 | 3
Not completed — Amputation - no longer eligible | 1 | 2
Not completed — Death | 1 | 0
Not completed — patient non-compliance | 3 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care | Total
Number analyzed (Participants) | 25 | 21 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 15 | 11 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 21 | 17 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 100% Re-epithelialization
Description: Primary outcome is number of participants with 100% epithelialization at 12 weeks of treatment as determined by investigator assessment of the ulcer and imaging.
Time Frame: 12 weeks
Population: Patients who completed 12 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care
Number analyzed (Participants) | 19 | 18
Participants | 14 | 6

2. Secondary Outcome: Change in Wound Area
Description: The difference in wound area from baseline to 100% re-epithelialization or week 12 will be summarized for each treatment group in each arm. Wound sizes were documented by the investigator at baseline to end of the treatment period for each participant.
Time Frame: 12 weeks
Population: Per protocol population including participants that completed the primary study endpoint/treatment period without withdrawal.
Measure: Mean (Standard Deviation); unit: Percentage of ulcer size decrease
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care
Number analyzed (Participants) | 19 | 18
Percentage of ulcer size decrease | 89.3 (20.8) | 62.9 (56.0)

3. Secondary Outcome: Time to Wound Closure
Description: The number of weeks from initial application of study treatment until complete re-epithelialization is first identified.
Time Frame: Up to 12 Weeks
Population: Per protocol population who completed the primary endpoint/treatment period without withdrawal
Measure: Mean (Standard Deviation); unit: Number of weeks
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care
Number analyzed (Participants) | 19 | 18
Number of weeks | 6.57 (3.0) | 7.0 (2.9)

4. Secondary Outcome: Number of Treatment Applications
Description: The number of study treatment applications including the initial application until 12 weeks or until complete re-epithelialization, whichever occurs first.
Time Frame: 12 weeks
Population: The per protocol population, which includes all patients that completed the primary endpoint/treatment period without withdrawal
Measure: Mean (Standard Deviation); unit: Average number of treatment applications
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care
Number analyzed (Participants) | 19 | 18
Average number of treatment applications | 6.8 (3.5) | 7.7 (3.5)

5. Other Pre Specified Outcome: Quality of Life - SF-36
Description: The survey will be completed at the day of initial application and at either 12 weeks or at complete re-epithelialization
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cost Effectiveness / Economic Model
Description: Cost data from the patient's treatment will be analyzed based on diagnoses, procedure and supply codes to determine cost efficacy and outcomes with the treatment pathway and related technology utilized during the course of care.
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Incidence of Adverse Events
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For each individual patient, data was collected over the 12 week treatment period or until complete re-epithelialization and 2 week follow up visit, up to a maximum of 14 weeks
Description: Adverse events were monitored starting at randomization and through the treatment period and 2 week follow up. Adverse events were not monitored during the 2 week run-in period
Arm/Group | Treatment With Synthetic Hybrid-Scale Fiber Matrix | Treatment With Standard of Care
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/25 | 2/21
Other Adverse Events (participants affected / at risk) | 6/25 | 2/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Synthetic Hybrid-Scale Fiber Matrix (N=25) | Treatment With Standard of Care (N=21)
Amputation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) — Loss or removal of a body part such as a toe.
Cerebral vascular accident (Cardiac disorders) | 1 (1) | 0 (0) — Stroke
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Synthetic Hybrid-Scale Fiber Matrix (N=25) | Treatment With Standard of Care (N=21)
Infection (Skin and subcutaneous tissue disorders) | 6 (25) | 2 (21) — The invasion and multiplication of microorganisms such as bacteria, viruses, and parasites that are not normally present within the body

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/84/NCT04918784/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT04918784/ICF_001.pdf